CLINICAL TRIAL: NCT03546998
Title: Incidence and Risk Factors for Development of Epidermoid Carcinoma in Esophageal Achalasia
Brief Title: Epidermoid Cancer Development in Esophageal Achalasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sandro Mattioli (Other)
Responsible Party: Sponsor-Investigator, Sandro Mattioli, Prof. Sandro Mattioli, University of Bologna
Organization: University of Bologna (Other)
Other Study IDs: Epidermoid cancer in achalasia
Record Dates: First submitted 2018-04-27; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Achalasia; Epidermoid Carcinoma
Keywords: epidermoid carcinoma; esophageal achalasia; risk factors
MeSH Terms: conditions — Esophageal Achalasia; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinical instrumental examinations — Achalasia patients were periodically submitted to clinical assessment, barium swallow (esophageal diameter and residual barium column were measured), endoscopy. Mucosal esophageal biopsies were taken in order to diagnose dysplasia or epidermoid carcinoma.

SUMMARY:
Esophageal achalasia is a precancerous condition for epidermoid carcinoma; incidence and risk factors for cancer development are not defined. Incidence and risk factors for epidermoid carcinoma development in achalasia patients were investigated.

DETAILED DESCRIPTION:
In order to define incidence and risk factors for epidermoid carcinoma 681 patients affected by esophageal achalasia observed since 1973 were followed up with no time limits according to a prospective follow-up protocol. The local institutional review board approved using the database from the division of thoracic surgery for research purposes. Clinical, radiological and endoscopic data of achalasia patients were collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary esophageal achalasia achieved by means of radiology, endoscopy and manometry

Exclusion Criteria:

* pseudoachalasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 681 patients admitted at the division of Clinica Chirurgica II of the University of Bologna from 1973 and undergone surgery, pneumatic dilations or medical therapy for esophageal achalasia.
Sampling Method: Non-Probability Sample
Enrollment: 681 (Estimated)
Dates: Start 1973-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of epidermoid carcinoma of the esophagus | 1 year
  Detection of epidermoid carcinoma of the esophagus by means of upper GI endoscopy

SECONDARY OUTCOMES:
Result of achalasia treatment by investigating dysphagia and gastro-esophageal reflux | 1 year
  Result of achalasia treatment assessed by means of semiquantitative grading scales of dysphagia and gastro-esophageal reflux

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli, MD, Principal Investigator — Department of Medical and Surgical Sciences-Alma Mater Studiorum-Università di Bologna
Locations (1):
- Division of Thoracic Surgery Maria Cecilia Hospital, Cotignola, RA, Italy

IPD SHARING:
Plan to Share IPD: No